CLINICAL TRIAL: NCT00585338
Title: Treatment of Vascular Lesions With a Tandem 532/1064 nm Laser
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of California, Irvine (Other)
Collaborators: Beckman Laser Institute University of California Irvine (Other)
Responsible Party: Principal Investigator, Beckman Laser Institute and Medical Center, Wangcun Jia, PhD., Research Scientist, University of California, Irvine
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20033086
Record Dates: First submitted 2007-12-18; First posted 2008-01-03 (Estimated); Last update posted 2022-10-20 (Actual); Status verified 2022-10

CONDITIONS: Vascular Lesion
Keywords: facial telangiectasia,; leg vein telangiectasia; Port Wine Stain birthmarks
MeSH Terms: interventions — Lasers

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Tandem 532/1064 nm Laser (Experimental): Treatment of Vascular LesionsWith a Tandem 532/1064 nm Laser
  Interventions: Device: Tandem 532/1064 nm Laser

INTERVENTIONS:
Device: Tandem 532/1064 nm Laser — Treatment of Vascular Lesions With a Tandem 532/1064 nm Laser
  Other Names: Treatment of Vascular Lesions

SUMMARY:
Dermatologists have for many years treated vascular lesions by a variety of modalities including cryosurgery, electrotherapy, dermabrasion and radiation.

It has been hypothesized that simultaneous delivery of these two wavelengths may provide safer, and in some cases more effective, vascular lesion removal.

The Tandem laser is capable of emitting multiple cryogen spurts intermittently with multiple 532/1064 nm laser pulses.This mode may reduce malformed blood vessels with a low incidence of long-term side effects.

DETAILED DESCRIPTION:
The researcher can determine the blanching of vascular lesions after Tandem laser with multiple 532/1064 nm laser pulses treatment.

The researcher will select one to four test sites spots for laser treatment. will be Different laser parameters can be used for each test site. The research will evaluate of the test sites at 6-12 weeks for bruising and blanching. Parameters of the test area with the greatest degree of blanching without adverse effects will be utilized for further treatment. If no test area is determined to have blanching without adverse effects, further test sites may be performed.

ELIGIBILITY:
Inclusion Criteria:

* Adult age 18 years and older
* Diagnosis of vascular lesion

Exclusion Criteria:

* Age <18
* Pregnancy
* History of cutaneous photosensitivity
* Any therapy to the proposed treatment sites within the previous two months
* Current participation in any other investigational drug or device evaluation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2007-12; Primary Completion 2010-10 (Actual); Study Completion 2010-10 (Actual)

PRIMARY OUTCOMES:
Laser treatment | 6 months
  Treatment of Vascular Lesions With a Tandem 532/1064 nm Laser

CONTACTS AND LOCATIONS:
Overall Officials: John S Nelson, M.D, PhD, Study Director — Beckman Laser Institute University of California Irvine; Wangcun Jia, PhD, Principal Investigator — Beckman Laser Institute University of California Irvine; Kristen Kelly, M.D, Principal Investigator — Beckman Laser Institute University of California Irvine
Locations (1):
- Beckman Laser Institute Medical and Surgical Clinic, Irvine, California, United States